CLINICAL TRIAL: NCT03100331
Title: Neuropsychological Outcomes of Internationally-Adopted Children Who Are Perinatally-Infected With Human Immunodeficiency Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-299
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: HIV/AIDS
Keywords: neuropsychological outcomes; HIV/AIDS; international adoption; perinatal infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm; all receive neuropsychological testing & follow-up (Experimental)
  Interventions: Other: Neuropsychological testing

INTERVENTIONS:
Other: Neuropsychological testing — Comprehensive neuropsychological assessment and implementation of appropriate support and resources.

SUMMARY:
Children who are perinatally-infected with HIV are extremely vulnerable to cognitive delays and psychiatric disease, and the risk for neuropsychiatric illness is compounded in children who are internationally-adopted and may have suffered trauma, abandonment, malnutrition and neglect. While cognitive and psychiatric issues have been described in HIV-infected children, and even more so in HIV-positive adults, there have been no reports on neuropsychiatric interventions that can improve cognitive and psychiatric states in this highly vulnerable population. Without these needed data, Pediatric HIV providers have not been able to advocate for optimal neuropsychiatric care in perinatally HIV-infected children, let alone those who has suffered the additional risk of being internationally adopted. In the proposed study, the investigators will report on the neuropsychological profiles and outcomes in a cohort of internationally-adopted, perinatally HIV-infected children between ages 6 to 16 years who have not previously undergone neuropsychological testing or treatment. Data obtained from this study will provide important contributions to the literature by building understanding of the complex needs of this population as well as guiding future intervention efforts. The investigators predict that intervention efforts aimed at helping educators understand the learning and cognitive challenges for many of our patients will guide targeted academic supports in the school setting and lead to gains in academic skills. The detailed information obtained during the comprehensive neuropsychological assessment and follow-up care will be shared with the child's key educators at school so that individualized educational strategies can be developed, while maintaining confidentiality regarding the child's HIV status.

ELIGIBILITY:
Inclusion Criteria:

* Perinatally infected with HIV, internationally adopted

Exclusion Criteria:

* Prior neuropsychological testing

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change in Rating scales of behavioral and social/emotional functioning | 24-36 months
  Parental reporting
Change in Score of Wechsler Intelligence Scale for Children - Fifth Edition | 24-36 months
Change in Score of Wechsler Individual Achievement Test - Third Edition | 24-36 months
Change in Score of Gordon Diagnostic System | 24-36 months
Change in Score of Grooved Pegboard | 24-36 months
Change in Score of Token Test for Children - Second Edition | 24-36 months
Change in Score of Wide Range Assessment of Memory and Learning - Second Edition | 24-36 months
Change in Score of Delis Kaplan Executive Function System: Selected Subtests | 24-36 months
Change in Score of Rey-Osterrieth Complex Figure Test | 24-36 months
Change in Score of Beery-Buktenica Developmental Test of Visual Motor Integration - Sixth Edition | 24-36 months
Change in Score of Peabody Picture Vocabulary Test - Fourth Edition | 24-36 months
Change in Score of Behavior Assessment System for Children - Second Edition: Self, Parent, and Teacher Reports | 24-36 months
Change in Score of Pediatric Sleep Questionnaire | 24-36 months

IPD SHARING:
Plan to Share IPD: Yes
We may share the data with future co-investigators at the NIH Peds HIV observational cohort study